CLINICAL TRIAL: NCT05183646
Title: A Pivotal Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of DMX-200 in Patients With Focal Segmental Glomerulosclerosis (FSGS) Who Are Receiving an Angiotensin II Receptor Blocker (ARB)
Brief Title: A Study of the Efficacy and Safety of DMX-200 in Patients With FSGS Who Are Receiving an ARB
Acronym: ACTION3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dimerix Bioscience Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMX-200-301; 2023-504597-37 (EudraCT Number)
Record Dates: First submitted 2021-11-29; First posted 2022-01-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: FSGS
Keywords: fsgs; focal segmental glomerulosclerosis; kidney disease
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Kidney Diseases | interventions — propagermanium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DMX-200 (repagermanium) (Experimental): Patients will receive 120 mg immediate release capsules of DMX-200 twice daily during the treatment period (104 weeks)
  OLE: Patients will receive 120 mg immediate release capsules of DMX-200 twice daily during the OLE period (108-212 weeks)
  Interventions: Drug: DMX-200
- Placebo (Placebo Comparator): Patients will receive 120 mg immediate release capsules of Placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DMX-200 — DMX-200 (repagermanium) is a C-C chemokine receptor type 2 (CCR2) inhibitor.
  Other Names: Repagermanium
  Arms: DMX-200 (repagermanium)
Drug: Placebo — Patients will receive 120 mg capsules of Placebo twice daily
  Arms: Placebo

SUMMARY:
DMX-200 (repagermanium) is a C-C chemokine receptor type 2 (CCR2) inhibitor that, when administered concurrently with an ARB, is designed to inhibit recruitment of monocytes implicated in the inflammatory chemokine environment of chronic disease. The purpose of this pivotal randomized double-blind study is to investigate the efficacy and safety of DMX-200 120 mg twice daily (BID) compared with placebo over a treatment period of 104 weeks in adult patients with FSGS who are being treated with an ARB. Given the rarity of the disease and the similarities between adults and pediatric patients with FSGS, Dimerix will also investigate the efficacy and safety of DMX 200 in adolescents aged 12 to 17 years. The double-blind period will be followed by an open-label extension (OLE) which aims to assess the long-term efficacy and safety of DMX 200 for up to 2 additional years.

DETAILED DESCRIPTION:
This is a pivotal Phase 3, multicenter, randomized, double-blind, placebo-controlled study of the efficacy and safety of DMX-200 in patients with FSGS. The duration of the double-blind period per patient is estimated to be maximum of 122 weeks, a Screening and Qualification period of between 6 and 14 weeks (including a 4 week period to complete the assessments required for Screening, Titration (if required, up to 4 weeks) and, 6-weeks of Stabilization, a 104-week Treatment period, and up to a 4-week off-treatment Follow-up period. The treatment duration of the OLE period per patient is estimated to be a minimum of 104 weeks (2 years) with a 4-week off-treatment Follow-up period. The total study duration (double-blind period and OLE combined) is currently estimated to be a minimum of 230 weeks.

ELIGIBILITY:
DOUBLE BLIND PERIOD

Inclusion Criteria:

1. Patients must be 12 to 80 years old
2. A diagnosis of primary FSGS, genetic FSGS, or FSGS of undetermined cause. Confirmed by kidney biopsy within 7 years of screening
3. Must be either receiving an ARB at the maximal tolerated dose or willing to transition
4. If taking corticosteroids, the dosage must be stable for ≥4 weeks prior to Screening and during Stabilization
5. If taking aldosterone inhibitors, mineralocorticoid receptor antagonists, direct renin inhibitors, sodium-glucose co-transporter-2 (SGLT2) inhibitors, or endothelin receptor antagonists (ERAs, including dual antagonists), the dose and regimen must be stable for ≥12 weeks prior to Screening and during Stabilization
6. Urine PCR >1.5 g/g (>169.5 mg/mmol) or 24-hour total protein >1.5 g/day based on 24-hour urine collection during Screening.
7. Estimated eGFR ≥25 and ≤120 mL/min/1.73 m2 at Screening for adults & eGFR ≥25mL/min/1.73 m2 for adolescent patients (<18 years)
8. Seated blood pressure ≤160/100 mm Hg (mean of 3 values) (patients ≥18 years of age) or between the 5th and 95th percentile for age, sex, and height (patients <18 years of age) at Screening
9. Body weight ≥35 kg (all patients) AND a body mass index (BMI) ≤40 kg/m2 (patients ≥18 years of age) or between the 5th and 98th percentile for age and sex (patients <18 years of age) at Screening.
10. A female patient is eligible to participate if she is not pregnant or planning to become pregnant during the study, not breastfeeding, and at least one of the following conditions applies:

    1. Is not of childbearing potential
    2. If of childbearing potential and beginning at menarche, agrees to use a highly effective method of contraception consistently during the treatment period.
11. A male patient with a female partner of childbearing potential is eligible to participate if he agrees to use acceptable contraception
12. A patient or parent/legal guardian (as appropriate) who is capable of giving signed informed consent, and where required, the patient is capable of providing assent.

Exclusion Criteria:

1. Has FSGS secondary to another condition.
2. Patients with nephrotic syndrome (>3.5 g/day proteinuria and serum albumin <30 g/L) who have not previously been treated with standard of care FSGS-directed therapies (including steroids).
3. History of type 1 diabetes mellitus, or uncontrolled type 2 diabetes mellitus (defined as glycated hemoglobin [HbA1c] >8% at Screening)
4. History of lymphoma, leukemia, or any active malignancy within the past 2 years (except for basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ that have been resected and with no evidence of metastatic disease).
5. Active clinically significant hepatobiliary disease.
6. Documented history of heart failure (New York Heart Association Class III/IV) or a major adverse cardiac event within 12 weeks prior to Screening.
7. Has a physical, medical, or psychological condition, that in the opinion of the Investigator, may interfere with the evaluation the study.
8. The patient has a history of alcohol or illicit drug use disorder within 1 year prior to Screening.
9. Had a prior organ transplant or stem cell transplant, with the exception of corneal transplant.
10. Positive screening assessment for viral hepatitis B surface antigen, or anti-hepatitis C virus (HCV) antibody AND positive HCV RNA, or human immunodeficiency virus 1 and 2.
11. Serum potassium levels >5.5 mmol/L at Screening.
12. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2 × upper limit of normal (ULN) at Screening.
13. Treatment with non-steroid immunosuppressant agents including biological drugs (e.g. rituximab), calcineurin inhibitors, cyclophosphamide, azathioprine, or mycophenolate mofetil within 12 weeks prior to Screening.
14. History of serious side effects or allergic response to an angiotensin II antagonist or has a known sensitivity to any components in the IP.
15. Unable to swallow oral medication.
16. Prior participation in any Dimerix-sponsored DMX-200 clinical study.
17. Participation in a clinical study with an investigational product (IP) within 28 days or 5 half-lives (whichever is longer) prior to Screening or plans to participate in another study during the course of this study.
18. Are study site personnel directly affiliated with this study and their immediate families

OLE PERIOD

Inclusion Criteria:

1. A patient or parent/legal guardian (as appropriate) who is capable of giving signed informed consent, and where required, the patient is capable of providing assent.
2. Patients who have completed participation in the double-blind period, including the Week 104 visit, and who may derive benefit from (continued) treatment with DMX-200, and/or continued follow-up
3. The patient received blinded Investigational Product throughout the duration of the double-blind period up to the Week 104 visit
4. The patient continues to meet the contraceptive requirements

Exclusion Criteria:

1. The patient has met the criteria for permanent IP discontinuation or study discontinuation
2. Any safety concerns identified during the double-blind period which, in the Investigator's opinion, may interfere with the patient's continued participation during the OLE period.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of DMX-200 in terms of urine protein/creatinine ratio (PCR) in patients with FSGS who are receiving an ARB. | Baseline to Week 35
  Percent change in urine PCR (based on 24-hour urine collection)
Evaluate the efficacy of DMX-200 in terms of estimated glomerular filtration rate (eGFR) slope in patients with FSGS who are receiving an ARB (Analysis at week 35 and Week 104). | Baseline to Week 104
  Slope of eGFR
OLE - Assess the long-term safety and tolerability of open-label treatment with DMX-200 in patients with FSGS who are receiving an ARB. | Double-blind baseline to Week 216
  Incidence and severity of treatment-related adverse events (AEs) and any adverse events of special interest (AESIs) and serious adverse events (SAEs) following long-term treatment with DMX-200.

SECONDARY OUTCOMES:
Evaluate the incidence and severity of AEs with treatment of DMX-200 in adult and adolescent patients with FSGS who are receiving an ARB. | Baseline to Week 104
  Incidence and severity of AEs and clinically significant changes following treatment with DMX-200 compared with placebo.
To evaluate the effect of DMX-200 on kidney function parameters including proteinuria in patients with FSGS who are receiving an ARB. | Baseline to Week 104
  Proportion of responders and non-responders following treatment with DMX-200 compared with placebo.
  Proportion of patients on treatment with DMX-200 compared with placebo that meet a composite endpoint of worsening in kidney function.
OLE - Assess the long-term efficacy of open-label treatment with DMX-200 in patients with FSGS who are receiving an ARB. | From Week 108 (Baseline) at each visit
  Slope of eGFR and percent change in urine PCR
OLE - Evaluate the long-term effect of open-label treatment with DMX-200 on kidney function parameters in patients with FSGS who are receiving an ARB. | Double blind baseline to Week 216
  Proportion of patients on treatment with DMX-200 that meet a composite endpoint of worsening in kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: David Fuller, Study Director — Dimerix Bioscience Pty Ltd
Locations (220):
- United States (54):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Kidney Disease and Hypertension Center, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Amicis Research Centre, Northridge, California
  - Northridge Clinical Research Inc., Northridge, California
  - Kaiser Permanente, Oakland, California
  - University of California Davis Health System, Sacramento, California
  - Scripps Health, San Diego, California
  - Stanford Hospital and Clinic, Stanford, California
  - University of Colorado Anschutz Medical Campus, Denver, Colorado
  - Denver Nephrology Research Division, Denver, Colorado
  - South Florida Nephrology Group, P.A., Coral Springs, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - CTR Oakwater LLC, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Georgia Nephrology, Lawrenceville, Georgia
  - Boise Kidney, Boise, Idaho
  - CARE Institute - Idaho Falls, Idaho Falls, Idaho
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Nephrology Associates of Northern Illinois and Indiana (NANI Research), Oak Brook, Illinois
  - University of Louisville, Louisville, Kentucky
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Intermed Consultants, Edina, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - CARE Institute - Nephrology & Hypertension Associates, Tupelo, Mississippi
  - Children's Mercy Research Institute, Kansas City, Missouri
  - Washington University, School of Medicine, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Kidney and Hypertension Center, Roseburg, Oregon
  - The Childrens Hospital of Philadelphia Kohls GI Nutrition and Diagnostic Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - South Carolina Clinical Research, North Charleston, South Carolina
  - Carolina Nephrology, PA, Spartanburg, South Carolina
  - Arlington Nephrology, Arlington, Texas
  - Nephrotex Research Group, Dallas, Texas
  - Renal Disease Research Institute, LLC - Dallas, Dallas, Texas
  - MedResearch, Inc, El Paso, Texas
  - University Texas Medical Branch, Galveston, Texas
  - Kaleidoscope Clinical Research, Houston, Texas
  - Clear Lake Specialties, Webster, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
- Argentina (8):
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Organizacion Medica de Investigacion (OMI), CABA
  - Centro Médico de Nutrición y Diabetes-CENUDIAB, Ciudad Autonoma Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital General de Agudos Dr. Cosme Argerich, Ciudad Autonoma Buenos Aires
  - Clinica Privada Velez Sarsfield, Córdoba
  - Clinica de Nefrologia Urologia y Enf. Cardiovasculares S.A., Santa Fe
- Australia (10):
  - Griffith University, Brisbane
  - Princess Alexandra Hospital, Brisbane
  - Austin Hospital, Melbourne
  - Monash Health, Melbourne
  - St Vincent's Hospital Melbourne, Melbourne
  - Western Health, Melbourne
  - John Hunter Hospital, Sydney
  - Liverpool Hospital, Sydney
  - Nepean Hospital, Sydney
  - Royal North Shore Hospital, Sydney
- Brazil (5):
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu
  - Hospital das Clínicas da Universidade Federal de Pernambuco, Recife
  - HUPE-UERJ - Hospital Universitário Pedro Ernesto - Universidade Estadual do Rio de Janeiro, Rio de Janeiro
  - Fundação Oswaldo Ramos - Hospital do Rim, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo
- China (19):
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Zhejiang University school of medicine, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Shandong Provincial Hospital, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai
  - Peking University Shenzhen Hospital, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - General Hospital of Ningxia Medical University, Yinchuan
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang
- Všeobecná fakultní nemocnice v Praze, Prague, Czechia
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Kolding Sygehus, Kolding
  - Odense University Hospital, Odense
- France (8):
  - Groupe Hospitalier Pellegrin, Bordeaux, Gironde
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble Hopital Nord, Grenoble
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Hopital de la Conception APHM, Marseille
  - Hopital Lapeyronie pt, Montpellier
  - Hôpital Necker Enfants Malades, Paris
  - CHU Saint Etienne Hôpital Nord, Saint-Priest-en-Jarez
- Germany (9):
  - Universitaetsklinikum Aachen AOeR, Aachen
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Zentrum fuer Nieren Hochdruck und Stoffwechselerkrankungen, Hanover
  - Universitaetsklinikum Schleswig Holstein - Campus Luebeck, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Nephrologischen Zentrum Villingen-Schwenningen, Villingen-Schwenningen
- Hong Kong (3):
  - Pok Oi Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong
- Italy (7):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale San Raffaele, Milan
  - Fondazione Salvatore Maugeri IRCCS, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Ospedale San Giovanni Bosco, Torino
- Japan (20):
  - Kasugai Municipal Hospital, Kasugai, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - NHO Chibahigashi National Hospital, Chiba, Chiba
  - Teikyo University Chiba Medical Center, Ichihara, Chiba
  - Kyushu University Hospital, Higashi, Fukuoka
  - Yokohama City University Hospital, Yokohama, Fukuura
  - Asahikawa Red Cross Hospital, Asahikawa, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara, Nara
  - Okayama University Hospital, Kitaku, Okayama-ken
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - The University of Osaka Hospital, Suita, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Tokushima University Hospital, Tokushima, Tokushima
  - Tokyo Women's Medical University Hospital, Tokyo, Tokyo
  - Nagoya University Hospital, Shōwaku, Tsurumaicho
  - Yamaguchi University Hospital, Ube, Yamaguchi
- Malaysia (7):
  - Hospital Serdang, Kajang, Selangor
  - Pusat Perubatan Universiti Kebangsaan Malaysia, Cheras
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Sunway Medical Centre, Petaling Jaya
- Mexico (5):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Servicios Hospitalarios De Mexico S A De C V, Chihuahua City
  - Neurociencias Estudios Clinicos, Culiacán
  - Hospital Civil Fray Antonio Alcalde, Guadalajara
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
- Portugal (9):
  - Centro Clinico Academico Braga, Associação (2CA-Braga), Braga
  - Centro Hospitalar de Lisboa Ocidental, E.P.E. Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar Universitario Lisboa Central E.P.E. Hospital Curry Cabral, Lisbon
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E. Hospital de Santa Maria, Lisbon
  - Hospital de Loures, E.P.E., Loures
  - Unidade Local de Saúde de São João, E.P.E, Porto
  - Centro Hospitalar de Setúbal, E.P.E., Hospital de São Bernardo, Setúbal
  - Unidade Local de Saude do Estuario Tejo E.P.E., Hospital Vila Franca de Xira, Vila Franca de Xira
  - Centro Hospitalar Vila Nova de Gaia/Espinho, E.P.E, Vila Nova de Gaia
- Spain (11):
  - Torrecárdenas University Hospital, Almería
  - Fundacion Puigvert, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
- Taiwan (8):
  - Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Shuangho Hospital Ministry of Health and Welfare, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
- Thailand (6):
  - Phramongkutklao Hospital, Bangkok
  - Siriraj Hospital, Bangkoknoi
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Khon Kaen
  - King Chulalongkorn Memorial Hospital, Pathum Wan
- Turkey (Türkiye) (8):
  - Ankara Training and Research Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Akdeniz University Faculty of Medicine, Antalya
  - Uludag University Medical Faculty, Bursa
  - Trakya University Medical Faculty, Edirne
  - Erciyes University Medical Faculty, Erciyes
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Kocaeli University Research and Application Hospital, Kocaeli
- United Kingdom (16):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Southmead Hospital, Bristol
  - Kent and Canterbury Hospital, Canterbury
  - St. Helier Hospital, Carshalton
  - University Hospital Coventry & Warwickshire, Coventry
  - Queen Elizabeth University Hospital, Glasgow
  - Leicester General Hospital, Leicester
  - Great Ormond Street Hospital for Children, London
  - Hammersmith Hospital, London
  - King's College Hospital, London
  - Royal Berkshire Hospital, Manchester
  - Royal Manchester Childrens Hospital, Manchester
  - Nottingham City Hospital, Nottingham
  - Salford Care Organisation, Salford
  - Northern General Hospital, Sheffield
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: No